CLINICAL TRIAL: NCT06217393
Title: Randomized Multicentre Open-label Study to Investigate the Non-inferiority of Itopride Hydrochloride 150mg Once Daily Versus Itopride Hydrochloride 50 mg Thrice Daily in Subjects With Functional (Non-ulcer) Dyspepsia or Chronic Gastritis
Brief Title: Trial of Itopride 150mg Once a Day Versus Itopride 50 mg Thrice a Day; in Patients With Functional Dyspepsia
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ITOP-322-0216
Record Dates: First submitted 2023-11-24; First posted 2024-01-22 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Functional Dyspepsia
Keywords: Functional Dyspepsia; gastrointestinal symptoms; gastric dysmotility; Bloating; Early satiety; postprandial fullness; upper abdominal pain; nausea and vomiting; anorexia; heartburn; chronic gastritis
MeSH Terms: conditions — Abdominal Pain; Nausea; Vomiting; Anorexia; Heartburn

STUDY DESIGN:
Intervention Model Description: This is a Phase 3, randomized, open-label, multicenter, parallel-group, active-controlled study to evaluate the non-inferiority efficacy of Itopride Hydrochloride 150mg extended release tablet ( administered once daily) compared to Itopride Hydrochloride 50 mg film coated tablets (administered TID) in subjects with gastrointestinal symptoms caused by gastric dysmotility and delayed gastric emptying, like sensation of bloating, early satiety, postprandial fullness, upper abdominal pain or discomfort, anorexia, heartburn, nausea and vomiting; functional (non-ulcer) dyspepsia or chronic gastritis. This study will enroll 564 subjects and the duration of subject participation will be approximately 11 weeks.
  Test group - Itopride Hydrochloride 150 mg extended release tablets once daily before one of the main meals (preferably the same meal throughout the treatment) Active Control group - Itopride Hydrochloride 50 mg film coated tablets 3 times daily before meals
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Itopride Hydrochloride 150 mg extended release tablets once daily before one of the main meals (Experimental): Test group - Itopride Hydrochloride 150 mg extended release tablets once daily before one of the main meals (preferably the same meal throughout the treatment)
  Interventions: Drug: Itopride Hydrochloride 150 mg extended release tablets
- Active Control group - Itopride Hydrochloride 50 mg film (Active Comparator)
  Interventions: Drug: Itopride Hydrochloride 50 mg film coated tablets

INTERVENTIONS:
Drug: Itopride Hydrochloride 150 mg extended release tablets — The intervention in the study is in form of test and active control groups- see details below • Test group - Itopride Hydrochloride 150 mg extended release tablets once daily before one of the main meals (preferably the same meal throughout the treatment)
  • Active Control group - Itopride Hydrochloride 50 mg film coated tablets 3 times daily before meals
  Arms: Itopride Hydrochloride 150 mg extended release tablets once daily before one of the main meals
Drug: Itopride Hydrochloride 50 mg film coated tablets — The intervention in the study is in form of test and active control groups- see details below • Test group - Itopride Hydrochloride 150 mg extended release tablets once daily before one of the main meals (preferably the same meal throughout the treatment)
  • Active Control group - Itopride Hydrochloride 50 mg film coated tablets 3 times daily before meals
  Arms: Active Control group - Itopride Hydrochloride 50 mg film

SUMMARY:
The study is conducted in patients with functional dyspepsia or chronic gastritis. The purpose of this study is to:

* assess whether the dose of Itopride Hydrochloride 150 mg extended release tablets, taken once daily has a similar effect on gastrointestinal symptoms caused by gastric dysmotility and delayed gastric emptying, like bloating sensation, early satiety, postprandial fullness, upper abdominal pain or discomfort, anorexia, heartburn, nausea and vomiting in functional (non-ulcer) dyspepsia or chronic gastritis, as Itopride Hydrochloride 50 mg film coated tablets administered thrice a day.
* investigate assessment of the treatment provided to each participant.
* monitor safety and tolerability of Itopride Hydrochloride 150 mg extended release tablets, taken once daily before one of the main meals (preferably same meal throughout the treatment) and Itopride Hydrochloride 50 mg film coated tablets thrice daily before meals.

DETAILED DESCRIPTION:
This is a muti-national study, in subjects with functional dyspepsia. The study will screen approximately 700 subjects and include 564 subjects (282 subjects in both arms Test and Active control arm) and the treatment will be given as follows.

* Test group - Itopride Hydrochloride 150 mg extended release tablets once daily before any of the main meals (preferably same meal throughout the treatment) OR
* Active Control group - Itopride Hydrochloride 50 mg film coated tablets thrice daily before meals Total study participation will include screening for two weeks, treatment duration of eight weeks and follow-up for one week after the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male and/or non-pregnant non-lactating female subjects aged above 18 years.
2. Subjects provided written informed consent and are willing to participate in the study.
3. Subjects with functional (non-ulcer) dyspepsia according to Rome IV criteria including postprandial distress syndrome (PDS) and with or without EPS (epigastric pain syndrome) with one or more of the following:

   * bothersome postprandial fullness,
   * bothersome early satiation
   * bothersome epigastric pain,
   * bothersome epigastric burning for at least 12 weeks in the preceding 6 months
4. No evidence of organic, systemic, metabolic or structural disease likely to explain symptoms - Subjects who have to undergone physical examination and lab tests (including white-cell and red-cell counts, measurement of fasting blood sugar and liver-function tests), abdominal ultrasonography, and upper GI endoscopy* in order to rule out structural cause for symptoms of FD.

   *history of upper GI endoscopy within 6 months prior to enrolment or at screening.
5. Baseline severity of at least moderate symptoms on LDQ (total score ≥ 9) at screening.
6. H. pylori negative documented test report within 3 months prior to enrolment or during screening.

Exclusion Criteria:

1. Known hypersensitivity to Itopride or any component of the formulation and to any other related drug.
2. Subject with history or presence of clinically relevant evidence of cardiovascular, neurological, gastrointestinal/hepatic, renal, psychiatric, respiratory, urogenital, hematologic/immunologic, HEENT (head, ears, eyes, nose, throat), dermatological/ connective tissue, musculoskeletal, metabolic/nutritional, drug hypersensitivity, allergy, endocrine, major surgery or other relevant disease as revealed by medical history requiring treatment which at investigator's discretion might interfere with the study.
3. Subjects who cannot be treated with Itopride in line with the prescribing information.
4. Subjects scheduled for surgery during the study.
5. Subjects with a history of difficulty in swallowing.
6. Subject requiring concomitant treatment with anticholinergic drugs, drugs with narrow therapeutic index, sustained release or enteric-coated formulations.
7. Subjects taking Acid release inhibitors (e.g. histamine-2-receptor [H2]- antagonists, proton pump inhibitors [PPI], or potassium-competitive acid blockers), antacids (e.g. aluminium- or magnesium hydroxide, sodium bicarbonate), gastric mucosa protectors (e.g. sucralfate, rebamipide).
8. Subject with history of unusual bleeding and family history for bleeding disorders.
9. Subjects with only reflux-related symptoms or who have predominantly reflux-related symptoms.
10. Subjects with esophagitis, Barrett's esophagus, erosions or peptic ulcer disease within one year prior to the study or Zollinger-Ellison Syndrome.
11. Dyspepsia that is exclusively relieved by defecation or associated with a change in stool frequency or stool form to exclude IBS.
12. Clinically significant ECG abnormalities.
13. Subjects treated with Itopride or any other gastroprokinetic within 4 weeks prior to screening.
14. Subjects who took non-steroidal anti-inflammatory drugs for more than 2 weeks prior to screening
15. Subjects with refractory FD1 (defined as FD presenting symptoms continuing for at least 6 months, unresponsive to at least two medical treatments such as PPIs, prokinetics, or H. pylori eradication) as per investigator's discretion
16. History of or known inflammatory bowel disease (IBD) or coeliac disease.
17. History of or known severe hepatic, renal, pancreatic, cardiac, metabolic, hematological or malignant disease or trimethylaminuria.
18. Subjects with changed smoking status within the last three months.
19. History of or known GI malignancy or ulcers associated to malignancy or any alarm features for GI malignancy, e.g. GI bleeding.
20. Subjects who do not meet the criteria stated in concomitant medication section.
21. Subjects with history of severe depression, anxiety or other psychological disorders.
22. Females with child-bearing potential must agree to use an acceptable method of contraception during the study.
23. Subjects in whom an increase in gastrointestinal motility could be harmful, e.g., (history of) gastrointestinal hemorrhage, mechanical obstruction or perforation.
24. Specific food intolerance which is relieved by diet modifications (e.g. lactose intolerance, celiac disease).
25. Subjects with confirmed IBS as per Rome IV criteria.
26. Current alcohol or drug abuse.
27. History of abdominal surgery except appendectomy, cholecystectomy or hysterectomy, tubal ligations, bladder slings or vasectomies.
28. Hepatic cirrhosis or abnormal liver laboratory findings (defined as >3xULN of ALT or AST).
29. Subjects under hemodialysis therapy or having advanced chronic kidney disease (defined as eGFR <60 mL/min).
30. History of or known congestive heart failure NYHA class III and IV, or any other uncontrolled chronic diseases, such as: uncontrolled hypertension (systolic/diastolic blood pressure ≥160/100 mmHg); uncontrolled diabetes (HbA1c >8%).
31. Subjects currently being known to be afflicted by serious infection(s), or any known severe illness(es) which are judged by the investigator could interfere with subjects' safety and/or study evaluation.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 564 (Actual)
Dates: Start 2024-02-28 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
To assess the comparable efficacy of Itopride Hydrochloride 150 mg extended release tablet (administered once daily) and Itopride Hydrochloride 50 mg film coated tablets (administered TID) after 8 weeks' treatment | 8 weeks
  Change in the overall severity of functional dyspepsia between baseline and week 8, as measured by the Leeds Dyspepsia Questionnaire (LDQ) severity score

SECONDARY OUTCOMES:
To assess the comparable efficacy of Itopride Hydrochloride 150mg extended release tablet (administered once daily) and Itopride Hydrochloride 50 mg film coated tablets (administered TID) after 4 weeks treatment. | 4 weeks
  Change in the overall severity of functional dyspepsia between baseline and week 4, as measured by the Leeds Dyspepsia Questionnaire (LDQ) severity score
To assess quality of life for the two treatment arms using Disease Specific Quality of Life (Short Form - Nepean Dyspepsia Index SF-NDI) at baseline and end of treatment | 8 weeks
  Disease Specific Quality of Life (Nepean Dyspepsia Index NDI) assessed at baseline and week 8
Assess the symptomatology (sensation of bloating, early satiety, abdominal pain or discomfort, epigastric pain, epigastric burning, anorexia, heartburn, nausea and vomiting) of the disease in both treatment arms after 4 and 8 weeks of treatment. | 8 weeks
  Change from baseline of NRS 11 score for symptoms (sensation of bloating, early satiety, postprandial fullness, upper abdominal pain or discomfort (epigastric pain, epigastric burning), anorexia (loss of appetite), heartburn, nausea and vomiting) after 4 and 8 weeks of treatment
Change in the overall severity of functional dyspepsia between baseline and week 4, as measured by the Leeds Dyspepsia Questionnaire (LDQ) severity score (range 0-40), where 0 is symptom free and 40 is severe dyspepsia | 8 weeks
  Responder analysis for adequate/satisfactory relief as assessed by LDQ and/or NRS 11

OTHER OUTCOMES:
Treatment acceptance by subjects using 5-point Likert scale at the end of the treatment; (1. Not at all satisfied, 2. Slightly satisfied, 3. Neutral, 4. Very satisfied, 5. Extremely satisfied.) | 8 weeks
  Treatment acceptance and ease of use assessed by subjects using 5-point Likert scale
To evaluate safety and tolerability in both treatment arms | 8 weeks
  To evaluate the safety and tolerability of the two treatments by assessing the following safety endpoints: Treatment emergent adverse events (TEAEs) as detected by physical examination, laboratory assessments and vital signs. For each unique treatment, treatment emergent AEs will be summarized per primary standard of care, per Highest Level Term by primary Standard of care and per preferred term by highest level term and primary standard of care.

CONTACTS AND LOCATIONS:
Overall Officials: Suntje Sander, Study Director — Abbott Laboratories GmbH
Locations (19):
- Armenia (4):
  - "Grigor Narekatsi" MC, CJSC, Yerevan
  - "Hera Med" LLC ("Medicus" Medical Center), Yerevan
  - "Institute of Surgery Mickaelyan" CJSC, Yerevan
  - Polyclinic N 12 Health State, CJSC, Yerevan
- Malaysia (4):
  - Hospital Sultanah Bahiyah, Alor Star
  - Queen Elizabeth Hospital, Kota Kinabalu
  - Pantai Hospital Kuala Lumpur, Kuala Lumpur
  - UMMC, Petaling Jaya
- Philippines (4):
  - Cebu Doctors University Hospital, Cebu City
  - Davao Doctors Hospital, Davao City
  - Health Cube Medical Clinics, Manila
  - GreenCity Medical Center, Pampanga
- Thailand (4):
  - Phramongkulklao Hospital, Bangkok
  - King Chulalongkorn Memorial, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai
  - Srinagarind Hospital, Khon Kaen
- Vietnam (3):
  - 103 Military Hospital, Hanoi
  - Bach Mai Hospital, Hanoi
  - Nguyen Tri Phuong Hospital, Ho Chi Minh City